CLINICAL TRIAL: NCT06201715
Title: Efficacy and Safety of Tofacitinib in Patients With Prurigo Nodularis: a Prospective, Observational Pilot Study
Brief Title: Efficacy and Safety of Tofacitinib in Patients With Prurigo Nodularis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20231186
Record Dates: First submitted 2024-01-02; First posted 2024-01-11 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2023-09

CONDITIONS: Prurigo Nodularis; Itch
MeSH Terms: conditions — Pruritus | interventions — tofacitinib

STUDY DESIGN:
Intervention Model Description: Tofacitinib, an oral pan-JAK inhibitor, mainly selective against JAK1 and JAK3.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tofacitinib (Experimental)
  Interventions: Drug: Tofacitinib 5 MG

INTERVENTIONS:
Drug: Tofacitinib 5 MG — 5mg tofacitinib tablet twice daily

SUMMARY:
The goal is to evaluate the efficacy and safety of tofacitinib in treating refractory prurigo nodularis.The main questions it aims to answer are

1. whether tofacitinib is effective in treating prurigo nodularis in the longpterm.
2. whether tofacitinib is safe in prurigo nodularis patients in the longpterm.

ELIGIBILITY:
Inclusion criteria:

1. age ≥18 years old;
2. patients diagnosed with PN with a duration of more than 6 months;
3. presence of at least 10 pruritic nodules;
4. a Worst Itch-Numeric Rating Scale (WI-NRS) score ≥7 one week before study;
5. a history of more than 2 weeks of ineffective topical glucocorticoid treatment or antihistamine therapy;
6. signed informed consent and cooperated with the follow up and complied the study protocol.

Exclusion criteria:

1. current used of biologic, systemic glucocorticoid or immunosuppressive agents; past used of jak inhibitors;
2. were pregnant or lactating;
3. abnormal findings for patients' complete blood count, liver functions, and kidney function tests;
4. presence of any infection or inflammatory; presence of active tumors or an increased risk of tumor complications；
5. systemic comorbidities that could interfere with or complicate study assessments.
6. those experiencing atopic dermatitis within 6 months were excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Investigator's global assessment | up to 12 weeks
  a 11-point scale ranging from -5 (obvious aggravation) to 5(marked improvement) points.
Prurigo Activity Score | up to 12 weeks
  The PAS is a 7-item questionnaire evaluating the type, distribution and size of pruriginous lesions, the representative body area and exact number of lesions, the activity in the terms of percentage of pruriginous lesions with excoriations/crusts on top and the percentage of healed pruriginous lesions, which is proved to be a useful tool to objectively measure PN patients over time.
Visual analogue scale (VAS) at week 12 | up to 12 weeks
  The VAS is a visual scale for itch on a horizontal 10-cm line, on which the left end is marked as "no itch" and the right end is marked "worst imaginable itch". We defined the average pruritus of the past 24 hours as VAS24h, average, and the worst and average pruritus of the past 4 weeks as VAS4w, worst and VAS4w, average.
Numeric rating scale at week 12 | up to 12 weeks
  The NRS is a similar tool for the measurement of itch ranging from 0 (no itch) to 10 (unbearable itch). Similarly, we defined the average and worst pruritus of the past 24 hours using NRS as NRS24h, average and NRS24h, worst.
Verbal rating scale (VRS) at week 12 | up to 12 weeks
  The VRS is a 5-point questionnaire that indicated different itching intensities as follows: 0=none; 1=mild; 2=moderate; 3=severe; 4= very severe. The VRS24h, average, VRS24h, worst and VRSevening represented 24-hour average, worst as well as average evening pruritus by VRS.
Dermatology Life Quality Index (DLQI) at week 12 | up to 12 weeks
  The DLQI is a questionnaire with scores ranging from 0 to 30. The total scores of 30 points represent the worst possible quality of life due to pruritus and a change of the score of ≥4 points is considered to be clinically important.
Itchy specific quality of life (Itchy QoL) at week 12 | up to 12 weeks
  The Itchy QoL includes 22 pruritus-specific items as follows: 6 symptoms, 7 functional limitation, and 9 emotions.

SECONDARY OUTCOMES:
the proportion of patients with reduction in WI-NRS by ≥4 points from baseline at week 12 and week 16. | up to 16 weeks
  WI-NRS represents Worst Itch-Numeric Rating Scale score

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are not publicly available due to the privacy of research participants but are available from the sponsor upon reasonable request.